CLINICAL TRIAL: NCT06895252
Title: Efficacy of Microbiome Manipulation Strategies (fecAL Microbial Transplantation OR Anti-inflammatory diEt OR Both) in Combination With 5-aminosalicylic Acid for Induction and Maintenance of Remission in Patients With Mild to Moderate tReatment Naive Active Ulcerative Colitis: a Multicentre Double-blind Factorial Randomized Controlled Trial(ALTER-UC)
Brief Title: A Study to Evaluate the Effect of Fecal Transplant and Dietary Changes on Disease Activity in Patients With Newly Diagnosed Active Ulcerative Colitis
Acronym: ALTER-UC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: All India Institute of Medical Sciences (Other)
Collaborators: Post Graduate Institute of Medical Education and Research, Chandigarh (Other); Institute of Medical Sciences of the Banaras Hindu University, India (Other); Dayanand Medical College and Hospital (Other); Indraprastha Institute of Information Technology Delhi (Other); Lisie Hospital (Other); Indian Council of Medical Research (Other Government); Lokmanya Tilak Municipal Medical College and Hospital (Other)
Responsible Party: Principal Investigator, Prof. Vineet Ahuja, Professor, All India Institute of Medical Sciences
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: AIIMSA2990/03.01.2025; EMDR/CARE/12/2023-0000572 (Other Grant/Funding Number: Indian Council of Medical Research)
Record Dates: First submitted 2025-03-03; First posted 2025-03-26 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Ulcerative Colitis (UC)
Keywords: factorial design; Randomized controlled trial; Fecal microbiota transplantation; Anti inflammatory diet; Ulcerative colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Sham transplantation with sham diet (Sham Comparator): 1. Oral placebo 1 BD for 3 days before first FMT
  2. Sham transplantation with instillation of clean water at 0, 2, and 6 weeks followed by (if treatment responder) - 8-weekly during maintenance between 10 to 42 weeks
  3. Sham diet for 48 weeks 4. 5-ASA for 48 weeks
  Interventions: Other: Sham transplantation; Other: Sham diet
- Fecal Microbiota Transplant(FMT) and Sham diet (Experimental): 1. Oral vancomycin 500 mg BD for 3 days before the first FMT.
  2. FMT via colonoscopy at 0, 2 and 6 weeks followed by (if treatment responder) 8 weekly during maintenance between 10 to 42 weeks
  3. Sham diet for 48 weeks 4. 5-ASA for 48 weeks
  Interventions: Other: Fecal Microbial Transplantation; Other: Sham diet
- Anti-inflammatory diet and sham transplantation (Experimental): 1. Oral placebo 1 BD for 3 days before first FMT
  2. Sham transplantation (clean water) via colonoscopy at 0, 2 and 6 weeks followed by (if treatment responder) 8 weekly during maintenance between 10 to 42 weeks
  3. Anti-inflammatory diet for 48 weeks 4. 5-ASA for 48 weeks
  Interventions: Other: Sham transplantation; Other: Anti inflammatory diet
- Fecal Microbiota Transplant(FMT) and Anti inflammatory diet (Experimental): 1. Oral vancomycin 500 mg BD for 3 days before the first FMT.
  2. FMT via colonoscopy at 0, 2 and 6 weeks followed by (if treatment responder) 8 weekly during maintenance between 10 to 42 weeks
  3. Anti-inflammatory diet for 48 weeks
  4. 5-ASA for 48 weeks
  Interventions: Other: Anti inflammatory diet; Other: Fecal Microbial Transplantation

INTERVENTIONS:
Other: Sham transplantation — Sham FMT will involve saline infusion via colonoscopy
  Arms: Anti-inflammatory diet and sham transplantation; Sham transplantation with sham diet
Other: Anti inflammatory diet — The modified diet plan will be given to each study participant
  Arms: Anti-inflammatory diet and sham transplantation; Fecal Microbiota Transplant(FMT) and Anti inflammatory diet
Other: Fecal Microbial Transplantation — This will involve colonoscopic instillation of fecal transplant
  Arms: Fecal Microbiota Transplant(FMT) and Anti inflammatory diet; Fecal Microbiota Transplant(FMT) and Sham diet
Other: Sham diet — Dietary counselling alone
  Arms: Fecal Microbiota Transplant(FMT) and Sham diet; Sham transplantation with sham diet

SUMMARY:
Ulcerative colitis (UC) is a chronic inflammatory condition affecting the colon and rectum, characterized by mucosal inflammation and symptomslike diarrhea, abdominal pain, and rectal bleeding. It is a subtype of inflammatory bowel disease (IBD) and results from a combination of genetic predisposition, environmental factors, and immune dysregulation. UC is associated with significant gut microbiota dysbiosis, marked by reduced beneficial bacteria and increased harmful taxa. With rising prevalence in developing countries like India, effective and accessible treatments remain a critical need. This multi-center randomized factorial double blind placebo controlled treat through trial will utilize a 2x 2 factorial design to randomize patients of mild to moderate (modified Mayo score 3-6) endoscopically active (Mayo endoscopic score: >1) treatment naÃive UC in 1:1:1:1 ratio to fecal microbiota transplantation (FMT) + anti-inflammatory diet (AID) +5-aminisalicylic acid (5-ASA) (Intervention, Group A) vs fecal microbiota transplantation + sham diet +5-aminisalicylic acid(Intervention, Group B) vs sham transplantation + anti-inflammatory diet +5-aminisalicylic acid(Intervention, Group C) vs sham transplantation

+ sham diet +5-aminisalicylic acid(Control, Group D). In the induction phase patients will receive FMT/sham transplantation at 0, 2 and 6 weeks along with AID/Sham diet and 5-ASA for 10 weeks. Outcome will be assessed at 10 weeks, Treatment failure will be out of trial. Patients with clinical response at 10 weeks will continue in the maintenance phase and will receive FMT/sham transplantation at 10, 18, 26, 34, and 42 weeks along with AID/Sham diet and 5-ASA till48 weeks. Outcome will be assessed at 48 weeks. Treatment failure will be out of trial. The primary efficacy outcome will evaluate fecal microbial transplantation or anti- inflammatory diet or combination of both vs placebo. The primary outcomes are proportion of patients having clinical remission and endoscopic response at week 10 and proportion of patients having clinical remission and endoscopic remission at week 48. Modified intention to treat analysis will be done and patients who receive at least 1 dose of intervention will be included for outcome assessment.

DETAILED DESCRIPTION:
This study is a multi-center, double-blind, 2 × 2 factorial, randomized sham-controlled trial designed to evaluate the effects of fecal microbiota transplantation (FMT) and dietary modification in treatment-naïve patients with mild to moderate active ulcerative colitis (UC). The trial consists of four treatment arms:

FMT + Anti-inflammatory Diet (AID) + 5-ASA (Group A) FMT + Sham Diet + 5-ASA (Group B) Sham Transplantation + AID + 5-ASA (Group C) Sham Transplantation + Sham Diet + 5-ASA (Group D) All groups receive 5-aminosalicylic acid (5-ASA) as the standard medical therapy.

Study Setting

The trial is conducted at six FMT centers across India, with one additional center dedicated to microbiome analysis:

AIIMS, New Delhi, India Dayanand Medical College, Ludhiana, India PGIMER, Chandigarh, India Lisie Hospital, Kochi, India IMS, BHU, Varanasi, India Lokmanya Tilak Municipal Medical College, Mumbai, India IIIT-Delhi, India (for microbiome analysis)

Intervention Details Fecal Microbiota Transplantation (FMT) Patients receive three FMT sessions (weeks 0, 2, 6) during induction and additional 8-weekly maintenance sessions (weeks 10, 18, 26, 34, 42) for responders.

FMT is delivered via colonoscopy; at week 0, it is instilled into the right colon/terminal ileum (post bowel preparation), while for maintenance sessions, it is instilled in the left colon without bowel preparation.

Each FMT dose is 50 g stool, freshly prepared within 4 hours of collection. Multiple donors are used to ensure microbiome diversity

Anti-Inflammatory Diet (AID) Patients assigned to AID receive a nutritionally tailored diet that promotes T-regulatory cell expansion, microbiome stability, and gut barrier integrity.

The diet excludes gluten-based grains, dairy products, and pro-inflammatory foods while including fermented foods, cruciferous vegetables, and polyphenols.

Patients are provided diet charts, receive dietary counseling, and are monitored via diet app named IBDNutricare.

Sham Interventions Sham FMT: Instead of donor stool, patients receive sterile water infusions via colonoscopy at the same time points as FMT.

Sham Diet: Patients receive dietary counselling without specific modifications

Randomization and Blinding Central randomization is conducted via REDCap. Block randomization will be done in which blocks of 8 will be created for the randomization. Further, stratified randomization will also be done in which <25% Proctitis involving Ulcerative Colitis patients.

Blinding:

Patients, investigators collecting clinical data, and those assessing endoscopic images are blinded. The endoscopist administering FMT and the dietitian providing dietary counseling are unblinded

Data Collection and Assessments Baseline Assessments (Week 0) Clinical Evaluation: Patient-reported outcomes (PRO-2), stool frequency, rectal bleeding assessments.

Laboratory Tests: Hemogram, renal/liver function, CRP, ESR, fecal calprotectin, and microbiome profiling.

Endoscopy: Mayo Endoscopic Score (MES) assessment with high-definition recordings.

Histology: Biopsy samples assessed using Robarts Histologic Index (RHI) and Distribution Chronicity and Activity (DCA) score

Follow-up Assessments Week 10 (Induction phase endpoint): Endoscopy, histology, laboratory tests. Week 48 (Maintenance phase endpoint): Same assessments as baseline. Microbiome Analysis: Fecal samples collected at baseline, 10 weeks, and 48 weeks for metagenomics and metabolomics

Safety Monitoring Adverse events graded using CTCAE criteria (Grade 1-5). Serious adverse events (SAEs) include hospitalization, disability, or life-threatening conditions

Data Management Data is collected using paper Case Report Forms (CRF's) and then data will be entered in REDCap.

Endoscopic images and videos are securely stored and centrally reviewed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with treatment-naive ulcerative colitis of any disease extent. Patients with proctitis will be limited to 25% of the entire pool of patients.
2. Mild to moderate endoscopically active disease (modified Mayo clinic score (mMS) 3-6, with Mayo endoscopic score greater than or equal to 2).
3. Aged between 18-75 years.
4. Patients giving consent for FMT.
5. Patients who agree to adhere to the diet schedule.
6. Patients on oral or topical ASA for less than 4 weeks.
7. Patients on oral steroids/ topical steroids for less than 1 week.
8. Infective colitis should be ruled out by histologic appearance of crypt architecture distortion/basal plasmacytosis, or two sigmoidoscopies, at least 7 days apart showing evidence of endoscopic activity.

Exclusion Criteria:

1. Patients with severe disease (mMS equal to 7-9)
2. Clinical signs of fulminant colitis or toxic megacolon
3. Presence of IBD-unclassified, microscopic colitis, ischemic colitis, infectious colitis, or clinical findings suggestive of Crohns Disease.
4. Patients who have been initiated on other therapies (biologicals or immunosuppressants (azathioprine/ 6-mercaptoprine/methotrexate)) for greater than 2 weeks
5. Patients requiring hospitalization
6. Pregnant or lactating women
7. Patients with current or recent history of clinically severe, progressive, or uncontrolled renal, hepatic, haematological, gastrointestinal, metabolic, endocrine, pulmonary, cardiac or neurological disease.
8. Positive assay or stool culture for pathogens (ova and parasite examination, bacteria) or positive test for Clostridioides difficile toxin at screening#
9. Patients infected with human immunodeficiency virus (HIV) # The patients with positive assay will be treated appropriately and tests will be repeated. Those with negative assay and persistent activity will be included in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2025-03-15 (Actual); Primary Completion 2027-03-15 (Estimated); Study Completion 2028-03-15 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients having clinical remission and endoscopic response at week 10 | 10 weeks
  Proportion of patients having-
  1. Clinical remission which is defined as the Modified Mayo Score (mMS) < 2 mMS- Full Title: Modified Mayo Score Range: 0 to 12 Higher Scores = Worse Outcome (A score of 0 represents no disease activity, and a score of 12 represents the most severe disease activity.)
  2. Endoscopic response which is defined as Mayo Endoscopic Score (MES) by 1 point MES- Full Title: Mayo Endoscopic Score Range: 0 to 4 Higher Scores = Worse Outcome (A score of 0 represents normal endoscopic findings, and a score of 4 represents severe mucosal damage.
Proportion of patients having clinical remission and endoscopic response at week 48 | 48 weeks
  Proportion of patients having-
  1. Clinical remission which is defined as the Modified Mayo Score (mMS) < 2 mMS- Full Title: Modified Mayo Score Range: 0 to 12 Higher Scores = Worse Outcome (A score of 0 represents no disease activity, and a score of 12 represents the most severe disease activity.)
  2. Endoscopic response which is defined as Mayo Endoscopic Score (MES) by 1 point MES- Full Title: Mayo Endoscopic Score Range: 0 to 4 Higher Scores = Worse Outcome (A score of 0 represents normal endoscopic findings, and a score of 4 represents severe mucosal damage.

SECONDARY OUTCOMES:
Proportion of patients having clinical response at week 10 | 10 weeks
  Proportion of patients having clinical response (Defined as a decrease from baseline in the mMS of greater than or equal to 2 points and at least a 30 percent reduction from baseline) mMS- Full Title: Modified Mayo Score Range: 0 to 12 Higher Scores = Worse Outcome (A score of 0 represents no disease activity, and a score of 12 represents the most severe disease activity.)
Proportion of patients having clinical remission at week 10 | 10 weeks
  Proportion of patients having clinical remission which is defined as an mMS of 0 to 2, including the following three components: 1) Stool frequency sub score = 0 (or = 1 with a ≥ 1-point decrease from baseline), 2) Rectal bleeding sub score = 0 3) Centrally read endoscopy sub score = 0 or 1 (score of 1 modified to exclude friability) mMS- Full Title: Modified Mayo Score Range: 0 to 12 Higher Scores = Worse Outcome (A score of 0 represents no disease activity, and a score of 12 represents the most severe disease activity.)
Proportion of Patients achieving Symptomatic Response at Week 10 | 10 weeks
  Proportion of Patients Achieving Symptomatic Response which is defined as Decrease from baseline ≥ 30% in composite Rectal Bleeding sub score and Stool Frequency sub score and a ≥ 1-point decrease from baseline in RB sub score or an absolute RB sub score ≤ 1)
  Stool Frequency Subscore:
  Range: 0 to 3 (typically; the exact range may vary depending on the scale used) Lower Scores = Better Outcome (A score of 0 indicates no stool frequency issues, while higher scores represent increasing frequency of stools, indicating worse disease activity.)
  Rectal Bleeding Subscore:
  Range: 0 to 3 (typically; range may vary depending on the version used) Lower Scores = Better Outcome (A score of 0 indicates no rectal bleeding, while higher scores represent increasing severity of rectal bleeding, indicating worse disease activity.)
Proportion of Patients achieving Symptomatic Remission at week 10 | 10 weeks
  Proportion of Patients achieving Symptomatic Remission which is defined as Stool Frequency subscore = 0 (or = 1 with a ≥ 1-point decrease from baseline) and Rectal Bleeding subscore = 0
  Stool Frequency Subscore:
  Range: 0 to 3 (typically; the exact range may vary depending on the scale used) Lower Scores = Better Outcome (A score of 0 indicates no stool frequency issues, while higher scores represent increasing frequency of stools, indicating worse disease activity.)
  Rectal Bleeding Subscore:
  Range: 0 to 3 (typically; range may vary depending on the version used) Lower Scores = Better Outcome (A score of 0 indicates no rectal bleeding, while higher scores represent increasing severity of rectal bleeding, indicating worse disease activity.)
Proportion of Patients Achieving Endoscopic Response at Week 10 | 10 weeks
  Proportion of Patients Achieving Endoscopic Response which is defined as decrease in Modified Endoscopic Score ≥1 points MES- Full Title: Mayo Endoscopic Score Range: 0 to 4 Higher Scores = Worse Outcome (A score of 0 represents normal endoscopic findings, and a score of 4 represents severe mucosal damage.
Proportion of Patients Achieving Endoscopic Remission at Week 10 | 10 weeks
  Proportion of Patients achieving Endoscopic Remission which is defined as Modified Endoscopy Score=0 MES- Full Title: Mayo Endoscopic Score Range: 0 to 4 Higher Scores = Worse Outcome (A score of 0 represents normal endoscopic findings, and a score of 4 represents severe mucosal damage.
Proportion of Patients Achieving Histologic Remission at Week 10 | 10 weeks
  Proportion of Patients Achieving Histologic Remission (Robarts histopathology index score <3 with lamina propria neutrophils score = 0 and neutrophil in epithelium score=0; DCA (Distribution/ chronicity/ activity) score, A=0)
  Robarts Histopathology Index (RHI):
  Full Title: Robarts Histopathology Index Range: 0 to 16 (varies depending on the specific version used, but typically it is in this range) Lower Scores = Better Outcome (A lower score indicates less histologic damage or inflammation.)
  Lamina Propria Neutrophils Score:
  Range: 0 to 3 Lower Scores = Better Outcome (A score of 0 indicates no neutrophils present, which is a sign of histologic remission.)
  Neutrophils in Epithelium Score:
  Range: 0 to 3 Lower Scores = Better Outcome (A score of 0 indicates no neutrophils in the epithelium, which is also a sign of histologic remission.)
  DCA Score:
  Full Title: Distribution/Chronicity/Activity Score Range: 0 to 3 Lower Scores = Better Outcome (score of 0 =no activity
Proportion of Patients Achieving Biomarker Remission at Week 10 | 10 weeks
  Proportion of Patients Achieving Biomarker Remission (Defined as fecal calprotectin ≤150 mcg/g)
Proportion of Patients Experiencing Adverse Events at Week 10 | 10 weeks
  Proportion of Patients experiencing Adverse events which will be assessed according to the Common Terminology Criteria for Adverse Events (CTCAE) and graded as follows: Grade 1: Mild symptoms (no intervention required). Grade 2: Moderate symptoms (non-operative intervention required). Grade 3: Severe symptoms (operative intervention required). Grade 4: Life-threatening consequences (urgent intervention required). Grade 5: Death.
Fecal Microbiome and Metabolite Signature at Week 10 | 10 weeks
  It involves combined analysis of the microorganisms (bacteria, viruses, fungi, etc.) and the small molecules (metabolites) present in a person's stool sample
Dynamics of microbiome engraftment at week 10 | 10 weeks
  It involves capturing donor-to-recipient microbiome transfer/shift at species and strain-level will be performed as an investigation of 'FMT events', where in each event will include triad of samples: the donor, the Pre-FMT and the Post-FMT sample from the recipient patient. Species-level donor-to-recipient shifts will be investigated by computing the Bray-Curtis and Kendall distances between all three sample-pairs of the triad.
  Kendall distances capture the variations and similarities amongst samples in terms of the relative hierarchical ranking of different taxa within a community, Bray-Curtis distances capture the differences in the abundances of different taxa across two communities. Both these distance measure-based approaches will be utilized the fraction of recipient microbiome that is modulated by the donor microbiome in terms of both composition and species-level hierarchy.
Proportion of patients having clinical response at week 48 | 48 weeks
  Proportion of patients having clinical response (Defined as a decrease from baseline in the mMS of greater than or equal to 2 points and at least a 30 percent reduction from baseline) mMS- Full Title: Modified Mayo Score Range: 0 to 12 Higher Scores = Worse Outcome (A score of 0 represents no disease activity, and a score of 12 represents the most severe disease activity.)
Proportion of patients having clinical remission at week 48 | 48 weeks
  Proportion of patients having clinical remission which is defined as an modified mayo score of 0 to 2, including the following three components: 1) Stool frequency sub score = 0 (or = 1 with a ≥ 1-point decrease from baseline), 2) Rectal bleeding sub score = 0 3) Centrally read endoscopy sub score = 0 or 1 (score of 1 modified to exclude friability) mMS- Full Title: Modified Mayo Score Range: 0 to 12 Higher Scores = Worse Outcome (A score of 0 represents no disease activity, and a score of 12 represents the most severe disease activity.)
Proportion of Patients Achieving Symptomatic Response at Week 48 | 48 weeks
  Proportion of Patients Achieving Symptomatic Response which is defined as Decrease from baseline ≥ 30% in composite Rectal Bleeding sub score and Stool Frequency sub score and a ≥ 1-point decrease from baseline in RB sub score or an absolute RB sub score ≤ 1) Stool Frequency Subscore: Range: 0 to 3 (typically; the exact range may vary depending on the scale used) Lower Scores = Better Outcome (A score of 0 indicates no stool frequency issues, while higher scores represent increasing frequency of stools, indicating worse disease activity.) Rectal Bleeding Subscore: Range: 0 to 3 (typically; range may vary depending on the version used) Lower Scores = Better Outcome (A score of 0 indicates no rectal bleeding, while higher scores represent increasing severity of rectal bleeding, indicating worse disease activity.)
Proportion of Patients achieving Symptomatic Remission at Week 48 | 48 weeks
  Proportion of Patients achieving Symptomatic Remission which is defined as Stool Frequency subscore = 0 (or = 1 with a ≥ 1-point decrease from baseline) and Rectal Bleeding subscore = 0 Stool Frequency Subscore: Range: 0 to 3 (typically; the exact range may vary depending on the scale used) Lower Scores = Better Outcome (A score of 0 indicates no stool frequency issues, while higher scores represent increasing frequency of stools, indicating worse disease activity.) Rectal Bleeding Subscore: Range: 0 to 3 (typically; range may vary depending on the version used) Lower Scores = Better Outcome (A score of 0 indicates no rectal bleeding, while higher scores represent increasing severity of rectal bleeding, indicating worse disease activity.)
Proportion of Patients achieving Endoscopic Response at Week 48 | 48 weeks
  Proportion of Patients Achieving Endoscopic Response which is defined as decrease in Modified Endoscopic Score ≥1 points MES- Full Title: Mayo Endoscopic Score Range: 0 to 4 Higher Scores = Worse Outcome (A score of 0 represents normal endoscopic findings, and a score of 4 represents severe mucosal damage.
Proportion of Patients achieving Endoscopic Remission at Week 48 | 48 weeks
  Proportion of Patients achieving Endoscopic Remission which is defined as Modified Endoscopy Score=0 MES- Full Title: Mayo Endoscopic Score Range: 0 to 4 Higher Scores = Worse Outcome (A score of 0 represents normal endoscopic findings, and a score of 4 represents severe mucosal damage.
Proportion of Patients achieving Histologic Remission at Week 48 | 48 weeks
  Proportion of Patients Achieving Histologic Remission (Robarts histopathology index score <3 with lamina propria neutrophils score = 0 and neutrophil in epithelium score=0; DCA (Distribution/ chronicity/ activity) score, A=0)
Proportion of Patients Achieving Biomarker Remission at Week 48 | 48 weeks
  Proportion of Patients Achieving Biomarker Remission (Defined as fecal calprotectin ≤150 mcg/g)
Fecal Microbiome and Metabolite Signature at Week 48 | 48 weeks
  It involves combined analysis of the microorganisms (bacteria, viruses, fungi, etc.) and the small molecules (metabolites) present in a person's stool sample
Dynamics of microbiome engraftment at week 48 | 48 weeks
  It involves capturing donor-to-recipient microbiome transfer/shift at species and strain-level will be performed as an investigation of 'FMT events', where in each event will include triad of samples: the donor, the Pre-FMT and the Post-FMT sample from the recipient patient. Species-level donor-to-recipient shifts will be investigated by computing the Bray-Curtis and Kendall distances between all three sample-pairs of the triad.
  Kendall distances capture the variations and similarities amongst samples in terms of the relative hierarchical ranking of different taxa within a community, Bray-Curtis distances capture the differences in the abundances of different taxa across two communities. Both these distance measure-based approaches will be utilized the fraction of recipient microbiome that is modulated by the donor microbiome in terms of both composition and species-level hierarchy.
Proportion of Patients Experiencing Adverse Events at Week 48 | 48 weeks
  Proportion of Patients experiencing Adverse events which will be assessed according to the Common Terminology Criteria for Adverse Events (CTCAE) and graded as follows: Grade 1: Mild symptoms (no intervention required). Grade 2: Moderate symptoms (non-operative intervention required). Grade 3: Severe symptoms (operative intervention required). Grade 4: Life-threatening consequences (urgent intervention required). Grade 5: Death
Proportion of patients having adverse events at week 6 | 6 weeks
  Proportion of Patients experiencing Adverse events which will be assessed according to the Common Terminology Criteria for Adverse Events (CTCAE) and graded as follows:
  Grade 1: Mild symptoms (no intervention required). Grade 2: Moderate symptoms (non-operative intervention required). Grade 3: Severe symptoms (operative intervention required). Grade 4: Life-threatening consequences (urgent intervention required). Grade 5: Death.
Proportion of patients having adverse events at week 26 | 26 weeks
  Proportion of Patients experiencing Adverse events which will be assessed according to the Common Terminology Criteria for Adverse Events (CTCAE) and graded as follows: Grade 1: Mild symptoms (no intervention required). Grade 2: Moderate symptoms (non-operative intervention required). Grade 3: Severe symptoms (operative intervention required). Grade 4: Life-threatening consequences (urgent intervention required). Grade 5: Death

CONTACTS AND LOCATIONS:
Locations (6):
- India (6):
  - Department of Gastroenterology, Lisie Hospital, Kochi, Kerala
  - Lokmanya Tilak Municipal General Hospital and Lokmanya Tilak Municipal Medical College, Sion, Mumbai, Maharashtra
  - Department of Gastroenterology and Human Nutrition, All India Institute of Medical Sciences, New Delhi, National Capital Territory of Delhi
  - Department of Gastroenterology, Dayanand Medical College, Ludhiana, Punjab
  - Department of Gastroentrology, Postgraduate Institute of Medical Education and Research, Chandigarh, Punjab/Haryana
  - Department of Gastroenterology, Institute of Medical Sciences, Banaras Hindu University, Varanasi, Uttar Pradesh

IPD SHARING:
Plan to Share IPD: No